CLINICAL TRIAL: NCT02382237
Title: Comparison of Tumor Glucose Metabolism Before and After Artificial Nutrition Assessed by F-FDG Petscan
Brief Title: Comparison of Tumor Glucose Metabolism Before and After Artificial Nutrition
Acronym: PETANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICM2013/31
Record Dates: First submitted 2014-02-04; First posted 2015-03-06 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer; Oesophageal Cancer
Keywords: denutrition in Head and Neck cancer or oesophageal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms | interventions — Injections; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/TDM (Other): Evaluation by PET/TDM at 2 times
  Interventions: Device: PET/TDM

INTERVENTIONS:
Device: PET/TDM — Evaluation of nutrition absorption by TEP/TDM
  Other Names: Parenteral or enteral nutrition

SUMMARY:
Evaluate the feasability to determine the difference of tumoral metabolism before and after artificial nutrition.

DETAILED DESCRIPTION:
Evaluation of the feasability to determine the difference of tumoral metabolism before and after artificial nutrition. This activity will be measured with TEP/TDM 18F-FDG

ELIGIBILITY:
Inclusion Criteria:

* VADS cancer or oesophageal cancer
* Evaluation by 18F-FDG PET
* denutrition with weight loss of 5%
* Artificial nutrition
* ECOG<2

Exclusion Criteria:

* Treatment by chemotherapy, surgery unless 2 months
* Treatment by radiotherapy unless 4 months
* Capillar glycemia >12mmol/l during the PET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
rate of Standardized Uptake Value (SUV) | 3 months
  The variation of the SUVmax is defined as the difference of the tumoral SUV max between the TEP1 and the TEP2

CONTACTS AND LOCATIONS:
Overall Officials: DESHAYES Emmanuel, Principal Investigator — ICM Co. Ltd.
Locations (1):
- ICM Val d'Aurelle, Montpellier, France